CLINICAL TRIAL: NCT05896930
Title: Phase 2 Trial to Evaluate the Early EBA, Safety and Tolerability of Amoxicillin/Clavulanate With or Without Meropenem, Ertapenem or Rifampicin in Adults With Newly Diagnosed, Smear-Positive Rifampicin-Susceptible Pulmonary Tuberculosis
Brief Title: Study to Evaluate EBA, Safety and Tolerability of Carbapenems in Adults With Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TASK Applied Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TASK 003
Record Dates: First submitted 2023-04-11; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Tuberculosis
Keywords: EBA; Intravenous Meropenem; Newly Diagnosed; Smear-Positive; Rifampicin-Susceptible; Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Meropenem; Ertapenem; Rifampin

STUDY DESIGN:
Intervention Model Description: This study will be a standard 14 day EBA design incorporating 2 groups with parallel treatment arms. This design allows comparison of the results of this study with similar prior studies of treatments for TB. No placebo treatment is included in this study - all participants will be given either active study treatment or Rifafour e275® control. The planned sample size is15 participants per treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Group 1 Arm 1 (Experimental): Meropenem 6g IV over 6 hours plus amoxicillin/CA
  Interventions: Drug: Meropenem 6g IV over 6 hours; Drug: Amoxicillin/CA twice daily
- Group 1 Arm 2 (Experimental): Ertapenem 1g IM plus amoxicillin/CA
  Interventions: Drug: Ertapenem 1g IM; Drug: Amoxicillin/CA twice daily
- Group 2 Arm 1 (Experimental): Meropenem 3g over 1 hour twice daily plus amoxicillin/CA
  Interventions: Drug: Meropenem 3g IV; Drug: Amoxicillin/CA twice daily
- Group 2 Arm 2 (Experimental): Ertapenem 1g IV plus amoxicillin/CA
  Interventions: Drug: Ertapenem 1g IV; Drug: Amoxicillin/CA twice daily
- Group 2 Arm 3 (Experimental): Amoxicillin; CA
  Interventions: Drug: Amoxicillin/CA twice daily
- Group 2 Arm 4 (Experimental): Rifampicin 35mg/kg plus amoxicillin/CA
  Interventions: Drug: Amoxicillin/CA twice daily; Drug: Rifampicin 35 mg/kg
- Group 2 Arm 5 (Experimental): Meropenem 6g or 4g IV over 60 minutes plus amoxicillin/CA
  Interventions: Drug: Meropenem 6g IV over 60 minutes; Drug: Meropenem 4g IV; Drug: Amoxicillin/CA once daily
- Group 1 (Active Comparator): Rifafour e-275
  Interventions: Drug: Rifafour e-275

INTERVENTIONS:
Drug: Meropenem 6g IV over 6 hours — Meropenem 6g intravenously over 6 hours once daily on days 1-14.
  Arms: Group 1 Arm 1
Drug: Ertapenem 1g IM — Ertapenem 1g intramuscularly once daily on days 1-14.
  Arms: Group 1 Arm 2
Drug: Meropenem 3g IV — Meropenem 3g intravenously twice daily over 60 minutes on days 1-14.
  Arms: Group 2 Arm 1
Drug: Ertapenem 1g IV — Ertapenem 1g intravenously once daily on days 1-14.
  Arms: Group 2 Arm 2
Drug: Amoxicillin/CA twice daily — Amoxicillin/CA 2 tablets x 1000mg/62.5mg orally 12-hourly on days 1-14.
  Arms: Group 1 Arm 1; Group 1 Arm 2; Group 2 Arm 1; Group 2 Arm 2; Group 2 Arm 3; Group 2 Arm 4
Drug: Rifampicin 35 mg/kg — Rifampicin 35 mg/kg once daily on days 1-14.
  Arms: Group 2 Arm 4
Drug: Meropenem 6g IV over 60 minutes — Meropenem 6g intravenously once daily over 60 minutes on days 1-14.
  Arms: Group 2 Arm 5
Drug: Rifafour e-275 — Rifafour e-275 will be supplied as fixed dose combination tablets and administered orally once daily for 14 days as The daily dose is dependent on the participants' weight as follows: 40 - 54kg: 3 tablets; 55 - 70kg: 4 tablets; 71kg and over: 5 tablets.
  Arms: Group 1
Drug: Meropenem 4g IV — Meropenem 4g intravenously once daily over 60 minutes on days 1-14.
  Arms: Group 2 Arm 5
Drug: Amoxicillin/CA once daily — Amoxicillin/CA 2 tablets x 1000mg/62.5mg orally once daily on days 1-14.
  Arms: Group 2 Arm 5

SUMMARY:
The goal of this single-center, open-labelled, clinical trial in two groups aims to proof that a specific group of antibiotics (carbapenems) can be used to treat pulmonary tuberculosis if it is combined with another antibiotic (amoxicillin/clavulanate). A total of 113 male or female participants (8 groups and 9 treatment regimens as group 8 was split into 2 groups of 4 participants receiving Rifafour e-275), aged between 18 and 65 years (inclusive), with newly diagnosed, smear-positive, pulmonary TB.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the 2-week bactericidal activity and pharmacokinetics of the following beta-lactam containing combinations with the aim to select the most active and implementable solution to be incorporated into a drug-resistant TB combination regimen:

* Once or twice daily meropenem administered intravenously in combination with once or twice daily oral amoxicillin/clavulanic acid;
* Once daily ertapenem administered intravenously and intramuscularly in combination with twice daily oral amoxicillin/clavulanic acid;
* Twice daily oral amoxicillin/clavulanic acid;
* Once daily rifampicin administered orally at highest currently established dosage of 35mg/kg in combination with twice daily oral amoxicillin/clavulanic acid.

A single-center, open-labeled, clinical trial in two groups. The treatments are:

Group 1:

1. Meropenem 6g intravenously once daily; plus amoxicillin/CA 2 x 1000mg/62.5mg orally 12-hourly on days 1-14.
2. Ertapenem 1g intramuscularly once daily; plus amoxicillin/CA 2 x 1000mg/62.5mg orally 12-hourly on days 1-14.

   Group 2:
3. Meropenem 3g intravenously twice daily; plus amoxicillin/CA 2 x 1000mg/62.5mg orally 12-hourly on days 1-14.
4. Ertapenem 1g intravenously once daily; plus amoxicillin/CA 2 x 1000mg/62.5mg orally 12-hourly on days 1-14.
5. Amoxicillin/CA 2 x 1000mg/62.5mg orally 12-hourly on days 1-14.
6. Rifampicin 35 mg/kg once daily; plus amoxicillin/CA 2 x 1000mg/62.5mg orally 12-hourly on days 1-14.
7. Meropenem 6g OR meropenem 4g intravenously once daily; plus amoxicillin/CA 2 x 1000mg/62.5mg orally once daily on days 1-14.

A total of 4 participants per group will receive standard first line TB treatment as per the South African TB guidelines (Rifafour e-275) and is included as a control for the EBA quantitative mycobacteriology and to evaluate whether HRZE gives similar EBA results to that demonstrated in prior studies with this combination. The mycobacteriology laboratory will remain blinded until closure of the EBA results. Enrollment into group 1 will be completed before enrollment into group 2 will start. After completion of enrollment into group 1, there will be an interim analysis while enrollment into group 2 is ongoing.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all trial-related procedures including HIV testing.
2. Male or female, aged between 18 and 65 years, inclusive.
3. Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
4. Newly diagnosed, previously untreated, rifampicin-susceptible pulmonary TB.
5. A chest X-ray picture which in the opinion of the Investigator is consistent with TB.
6. Sputum positive on direct microscopy for acid-fast bacilli on at least one sputum sample (at least 1+ on the IUATLD/WHO scale).
7. Ability to produce an adequate volume of sputum as estimated from an overnight sputum collection sample (estimated 10 ml or more).
8. Be of non-childbearing potential or using effective methods of birth control, as defined below:

Non-childbearing potential:

1. Participant - not heterosexually active or practicing sexual abstinence; or
2. Female participant/sexual partner - bilateral oophorectomy, bilateral tubal ligation and/or hysterectomy or has been postmenopausal with a history of no menses for at least 12 consecutive months; or
3. Male participant/sexual partner - vasectomised or has had a bilateral orchidectomy minimally three month prior to screening;

Effective birth control methods:

1. Double barrier method which can include a male condom, diaphragm, cervical cap, or female condom (male and female condoms should not be used together); or
2. Barrier method combined with hormone-based contraceptives or an intra-uterine device for the female partner; and are willing to continue practicing birth control methods throughout participation in the study until Visit 19 (day 28).

(Note: hormone-based contraception alone may not be reliable when taking IP; therefore, hormone-based contraceptives alone cannot be used by female participants to prevent pregnancy).

Exclusion Criteria:

1. Evidence of clinically significant conditions or findings, other than the indication being studied, particularly epilepsy, that might compromise safety or the interpretation of trial endpoints, per discretion of the Investigator.
2. Poor general condition where any delay in treatment cannot be tolerated per discretion of the Investigator.
3. A history of TB less than 3 years ago.
4. Clinically significant evidence of extrathoracic TB (miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the Investigator.
5. History of allergy to any of the trial IP/s or related substances i.e. β-lactams and penicillin, as confirmed by the clinical judgement of the Investigator.
6. Known or suspected, current or history of within the past 2 years, alcohol or drug abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the participant.
7. HIV infected participants.
8. Having participated in other clinical studies with investigational agents within 8 weeks prior to trial start.
9. Female participant who is pregnant, breast-feeding, or planning to conceive a child within the anticipated period of participating in the trial. Male participant planning to conceive a child within the anticipated period of participating in the trial.
10. Subjects with diabetes (Type 1 or 2), point of care HbA1c above 6.5, or random glucose over 11.1 mmol/L.
11. Hypersensitivity to local anaesthesia of amide type.
12. Treatment received with any drug active against MTB (including but not limited to isoniazid, ethambutol, amikacin, cycloserine, fluoroquinolones, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, thioamides, metronidazole), or with immunosuppressive medications such as TNF-alpha inhibitors or systemic or inhaled corticosteroids, within 2 weeks prior to screening
13. Participants with the following toxicities at screening as defined by the enhanced CTCEA toxicity table

    1. creatinine grade 2 or greater (>1.5 times upper limit of normal [ULN]);
    2. haemoglobin <7.5 g/dL;
    3. platelets grade 2 or greater (under 50x109 cells/L);
    4. serum potassium grade 2 or greater (<3.0 mEq/L);
    5. aspartate aminotransferase (AST) grade 3 (≥3.0 x ULN) to be excluded;
    6. alanine aminotransferase (ALT) grade 3 (≥3.0 x ULN) to be excluded;
    7. APTT grade 3
    8. INR grade 3
    9. Total white cell count grade 3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Early bactericidal activity by change in logCFU over 14 days | 14 days
  The EBACFU(0-14) as determined by the rate of change in logCFU (colony forming units) per ml sputum over the period Day 0 to Day 14 which will be summarised and described with a statistical model as an estimated average decrease per day for patients in each group.
Early bactericidal activity by change in time-to-positivity over 14 days | 14 days
  The EBATTP(0-14) as determined by the percentage rate of change in TTP (time to positivity) per ml sputum over the period Day 0 to Day 14, which will be summarised and described with a statistical model as an estimated average increase per day for patients in each group.

SECONDARY OUTCOMES:
Early bactericidal activity by change in logCFU and TTP per ml over 0-2 days, 0-7 days, and 2-14 days | 0-2 days, 0-7 days, 2-14 days
  Drug activity with CFU or TTP over different treatment periods such as 0-2 days, 0-7 days, and 2-14 days as indicated, for cross-comparison with other published data.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Andreas H Diacon, MD, PhD, Principal Investigator — TASK
Locations (1):
- TASK Clinical Research Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT05896930/Prot_SAP_000.pdf